CLINICAL TRIAL: NCT06646705
Title: Biochemical Evaluation of the Effect of Orthodontic Treatment with Aligner on Periodontal Parameters and OPG and RANKL Salivary Values
Brief Title: Biochemical Evaluation of Periodontal Effects of Orthodontic Treatment with Aligners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Burçin Akan, Doç. Dr., Izmir Katip Celebi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-GAP-DİŞF-0006
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Aligner Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aligner (Experimental): Full-mouth clinical periodontal measurements recorded and saliva obtained
  Interventions: Diagnostic Test: Saliva obtaining

INTERVENTIONS:
Diagnostic Test: Saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.

SUMMARY:
The aim of this study was to determine the effect of orthodontic treatment with aligner on changes in osteoprotegerin (OPG) and receptor activator of NF-κB ligand (RANKL) levels in saliva samples and to investigate the possible relationship between periodontal clinical parameters. Materials and Methods: A total of 25 (n=25) saliva samples were taken from systemically healthy non-smoking individuals who were planned to receive orthodontic treatment with aligner before treatment. Whole mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were also recorded and repeated at 1 and 3 months. Enzyme-linked immunosorbent assay (ELISA) was used to determine OPG and RANKL levels in biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (The determination of healthy volunteers will be based on the statements of the patients in the anamnesis. No additional examinations will be made.)
* Must receive orthodontic treatment with aligners and must have accepted the treatment
* Non-smoker
* No medication for continuous use
* Those who have not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 6 months.
* Not in pregnancy or lactation period.

Exclusion Criteria:

* Any oral or systemic disease
* Regularly using a systemic medication
* During pregnancy or lactation
* Received periodontal treatment within the last 6 months.
* Those who received antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months
* Smokers are not included in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The total amount of OPG in saliva | 24 hours after taking the clinical measurements
  The total amount of osteoprotegerin in saliva

SECONDARY OUTCOMES:
The total amount of RANKL in saliva | 24 hours after taking the clinical measurements
  The total amount of receptor activator of NF-κB ligand in saliva

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Çelebi University Faculty of Dentistry, Izmir, Cigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF